CLINICAL TRIAL: NCT02327403
Title: The B7-1 Study": Belatacept Conversion in Proteinuric Renal Transplant Recipients: an Interventional Multi-Center Trial
Brief Title: Belatacept Conversion in Proteinuric Kidney Transplant Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Leonardo V. Riella, MD PhD, Assistant Professor of Medicine, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015P000154
Record Dates: First submitted 2014-12-22; First posted 2014-12-30 (Estimated); Results first posted 2022-11-09 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-10

CONDITIONS: Proteinuria
Keywords: Proteinuria; Kidney transplantation; Allograft dysfunction; B7-1; Belatacept
MeSH Terms: conditions — Proteinuria | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Proteinuric Kidney Transplant Recipients (Experimental): Belatacept conversion
  Interventions: Drug: Belatacept

INTERVENTIONS:
Drug: Belatacept — Conversion from calcineurin-inhibitor to Belatacept maintenance immunosuppression.

SUMMARY:
Background: Proteinuria develops in about 30% of kidney transplant recipients and is a strong predictor of graft loss. The amount of proteinuria has a direct correlation with the risk of graft failure. Novel therapies are urgently needed to reduce proteinuria and prevent graft loss in transplant recipients, since ACE inhibitors carry a number of limitations in the transplant setting, including significant reduction in renal function, anemia and hyperkalemia.

Preliminary data: B7-1 is expressed at significant levels in about 10% of kidney allograft biopsies with predominance in patients with proteinuria.

Hypothesis: We hypothesize that B7-1 targeting therapy may reduce proteinuria and improve graft survival in proteinuric transplant recipients that have B7-1 staining on allografts. In addition, the absence of CNI nephrotoxicity and the potential protective effect of Belatacept on DSA production may be of benefit in this subset of transplant patients.

Objectives:

Primary: Determine the effect of Belatacept conversion in reducing proteinuria by 25% at 12 months in renal transplant recipients (≥1gram/d) that are either B7-1-positive or negative on kidney biopsy.

Secondary: Assess the effect of Belatacept conversion in the percent change of renal function from baseline to 12 months; donor-specific anti-HLA antibodies presence and intensity (MFI); correlation of B7-1 positivity on immunofluorescence on biopsy with B7-1-expression in urine extracellular vesicles; adverse events; acute rejection episodes; blood pressure control; new onset diabetes; hyperlipidemia; graft survival; and patient survival.

DETAILED DESCRIPTION:
A total of 36 patients will be recruited.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult kidney transplant recipients older than 18 years old
2. eGFR ≥30 ml/min
3. ≥6 months after transplantation
4. Proteinuria ≥1 gram/day in spot urine protein/creatinine ratio
5. Ability to provide written informed consent for the study.
6. Maintenance immunosuppression of CNI (cyclosporine or tacrolimus), antiproliferative agent (azathioprine, MMF or MPA) with either steroids or not.

Exclusion Criteria:

1. Age <18 years
2. eGFR<30 ml/min
3. active acute cellular rejection (ACR; higher than borderline) or ACR in the previous 6 months; active acute antibody-mediated rejection
4. recurrent FSGS
5. EBV IgG negative
6. patient on mTOR inhibitor (e.g. Everolimus, Sirolimus)
7. patient only on CNI (cyclosporine or tacrolimus) and steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo V Riella, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Belatacept Conversion: Kidney Transplant recipients with proteinuria who converted their immunosuppression from CNI to belatacept-based maintenance therapy
Period: Overall Study
Arm/Group | Belatacept Conversion
Started | 15
Completed | 13
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Belatacept Conversion: Belatacept: Conversion from calcineurin-inhibitor to Belatacept maintenance immunosuppression.
Arm/Group | Belatacept Conversion
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Black | 3
  Ethnicity: White | 7
  Ethnicity: Asian | 2
  Ethnicity: Hispanic | 3
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Proteinuria by 25%
Description: Change in proteinuria by 25%: daily proteinuria is estimated by spot urine protein (mg/dL) to creatinine (mg/dL) ratio at baseline (before the belatacept conversion) and post-conversion 12 months; and interval % change was calculated by getting the ratio of difference between the two time points to the baseline value.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Belatacept Conversion
Number analyzed (Participants) | 13
Participants | 8

2. Secondary Outcome: Change in Renal Function (eGFR in mL/Min/1.73 m^2)
Time Frame: from baseline to 12 months
Measure: Mean (Standard Deviation); unit: mL/min/1.73m2
Arm/Group | Belatacept Conversion
Number analyzed (Participants) | 13
mL/min/1.73m2
  Baseline | 45.8 (13.3)
  12 Months | 45.1 (12.7)

3. Secondary Outcome: Acute Rejection Episodes
Description: Acute rejection episodes [Time Frame: 12 months]: Number of biopsy-proven rejection episodes from belatacept conversion to post-conversion 12 months.
Time Frame: 12 months
Measure: Number; unit: episodes
Arm/Group | Belatacept Conversion
Number analyzed (Participants) | 13
episodes | 0

4. Secondary Outcome: Change in Blood Pressure Measurement (mm Hg)
Description: Change in Blood pressure measurement (mm Hg) [Time Frame: 12 months]: The mmHg difference in systolic and diastolic blood pressures between the baseline (pre-belatacept conversion) and post-conversion 12 months is assessed. Blood pressure measurement done at the office visits at baseline and 12 months after at least 5 minutes of resting.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Belatacept Conversion
Number analyzed (Participants) | 13
mmHg
  Baseline (Systolic) | 140 (11)
  Baseline (Diastolic) | 76 (6)
  12 Months (Systolic) | 129 (16)
  12 Months (Diastolic) | 72 (9)

5. Secondary Outcome: Change in Fasting Glucose
Description: New onset diabetes [Time Frame: 12 months]: Number of new onset diabetes per American Diabetes Association 2015 Criteria from belatacept conversion to post-conversion 12 months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Belatacept Conversion
Number analyzed (Participants) | 13
mg/dL
  Baseline | 119 (37)
  12 Months | 124 (62)

6. Secondary Outcome: Hyperlipidemia
Description: Hyperlipidemia [ Time Frame: 12 months]: Changes (mg/dL) in serum total cholesterol, LDL, HDL, and triglyceride levels from pre-belatacept conversion to post-conversion 12 months.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Belatacept Conversion
Number analyzed (Participants) | 13
mg/dL
  Baseline Total Cholesterol | 177 (49)
  12 Month Total Cholesterol | 171 (49)

7. Secondary Outcome: Graft Survival
Description: Graft survival [Time Frame: 12 months]: Number of patients who developed end stage kidney disease and required kidney replacement therapy within 12 months post-belatacept conversion.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Belatacept Conversion
Number analyzed (Participants) | 13
Participants | 13

8. Secondary Outcome: Patient Survival
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Belatacept Conversion
Number analyzed (Participants) | 15
Participants | 14

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Belatacept Conversion
All-Cause Mortality (participants affected / at risk) | 1/15
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 9/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belatacept Conversion (N=15)
Cardiac Arrest (Cardiac disorders) | 1 (1) — Cardiac arrest leading to death
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belatacept Conversion (N=15)
Pneumonia (Infections and infestations) | 2 (2)
Shingles (Infections and infestations) | 1 (1)
MRSA Cellulitis with Abscess (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) — Due to interstitial inflammation
Syncope (Nervous system disorders) | 1 (1)
Basal Cell Carcinoma (Skin and subcutaneous tissue disorders) | 1 (1)
Recurrence of Bladder Tumor (Renal and urinary disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-09): https://cdn.clinicaltrials.gov/large-docs/03/NCT02327403/Prot_SAP_000.pdf